Psychological Therapies Service
Golden Jubilee National Hospital
Agamemnon Street
Clydebank
G81 4DY
07970 496554
Gjnh.psychology@gjnh.scot.nhs.uk





## **CONSENT FORM**

## **Participant Number:**

Title of Project: The Relationship Between Interoception and Psychological Outcomes: A Mind-Body Intervention in Patients with Pulmonary Hypertension

Name of Researcher: Derick Moore

| | | Please initial box |
|---|---|---|
| 1. | I confirm that I have read the information sheet dated (version) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | |
| 3. | I understand that the project is a randomised control trial, which means that I may be randomised to the waitlist group that does not receive the treatment immediately but I will still be asked to complete a series of questionnaires. I understand that I will be contacted shortly after the first group has completed treatment to begin the intervention myself. | |
| 4. | I agree to provide my contact details for the purpose of the study and for Derick Moore (lead researcher) to contact me at the end of the intervention to complete a series of questionnaires. | |
| 5. | I understand that relevant sections of my medical notes and data collected during the study may be looked at by researchers from the regulatory authorities or from the NHS board, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | |

| 6. | I understand that anonymised information collected as part of this study may be used to support other research in the future and may be shared with other researchers. |
|---|---|
| 7. | I understand that if for any reason I lose my ability to make decisions throughout the duration of this study, the researchers will retain my personal data and continue to use this in a confidential manner, with the purpose for which my consent was originally sought. |
| 8. | I understand that any identifiable information collected will be deleted within three months of the study completion. |
| 9. | I understand that my General Practitioner (GP) will be informed of my participation in the study. |
| 10. | I understand that if I say something that indicates risk to myself or others, the researchers will have to pass this information on to relevant staff. |
| 11. | I agree to take part in the above study. I am aware, however, that I may not be included in the study if I do not meet the study inclusion criteria as part of the screening process. |
| 12. | I would like to receive a summary of the study findings once complete: YES NO |

Signature

Signature

Interoceptive Based Intervention in Pulmonary Hypertension: Consent form (Version 3 30/04/24). IRAS ID: 337496

Date

Date

Name of Participant

Name of Researcher

Derick Moore